CLINICAL TRIAL: NCT06365125
Title: Enhancing Computer-delivered Approaches to Reduce Heavy/Hazardous Alcohol Use Among College Students
Brief Title: College Student Daily Life and Alcohol Use Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 7313E
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Drinking, College; Drinking Heavy
Keywords: heavy alcohol use; college student; brief alcohol intervention
MeSH Terms: conditions — Alcohol Drinking in College

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Assessment Only (No Intervention): Assessment only condition, no intervention material delivered to this group
- Intervention (BAI) Only (Active Comparator): Only the brief alcohol intervention, eCHECKUP TO GO, is administered to this group
  Interventions: Behavioral: eCHECKUP TO GO
- Enhanced Intervention (Experimental): Brief alcohol intervention, eCHECKUP TO GO, + 4 weeks of text messaging boosters (Monday, Thursday-Sunday)
  Interventions: Behavioral: eCHECKUP TO GO; Behavioral: Text messaging boosters

INTERVENTIONS:
Behavioral: eCHECKUP TO GO — Single session, web-based intervention for college students aimed at increasing awareness of consequences related to heavy alcohol use and increase motivation to modify one's alcohol use.
  Other Names: eCHUG (former name)
  Arms: Enhanced Intervention; Intervention (BAI) Only
Behavioral: Text messaging boosters — Text messages sent a few times per week following completion of eCHECKUP TO GO to reinforce concepts and assist with goal setting and goal attainment in everyday life
  Arms: Enhanced Intervention

SUMMARY:
Heavy alcohol use among college students is associated with a range of negative consequences. However, college students rarely seek resources or treatment to change their alcohol use. Brief alcohol interventions (BAIs) have been developed as an alternative method to address heavy alcohol use among college students and show promise in reducing hazardous alcohol use in college students. Despite the established efficacy of BAIs, effects are often small and short-lived, and additional research is needed to investigate how BAIs can become more efficacious and endure for longer periods of time, particularly for computer-delivered interventions to improve accessibility and scalability of these interventions to a wider range of college students. Boosters or adjunctive components to BAIs have been suggested as a method to enhance the magnitude and duration of intervention effects. However, there remains a need to identify and test booster approaches that are both appealing and engaging to college students and effective in reducing heavy/hazardous alcohol use above and beyond the magnitude and duration seen by BAIs alone. The purpose of the study is to develop and test a novel, text-messaging booster as an adjunct to a current, evidence-based brief intervention, eCHECKUP TO GO, aimed at reducing college student heavy/hazardous alcohol use. Participants will complete baseline measures and will then be randomized to 1 of 3 conditions, stratified by sex at birth: 1) assessment only, 2) BAI only, and 3) Enhanced Intervention (BAI + four weeks of text messaging boosters). It is hypothesized that those randomized to the enhanced intervention condition will show a greater reduction in heavy/hazardous alcohol use at 3-month follow-up compared to the BAI and assessment only groups.

ELIGIBILITY:
Inclusion Criteria:

* 1) Ages 18-30; 2) report at least 2 heavy drinking episodes in the past month; 3) be enrolled in an undergraduate degree program; 4) own a smartphone with capability to run smartphone application

Exclusion Criteria:

* 1) current or past-year treatment (counseling or medication) for alcohol or drug use, 2) history of delirium tremens and/or seizures as a result of alcohol withdrawal, and 3) a lifetime diagnosis of either bipolar disorder or schizophrenia

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 129 (Estimated)
Dates: Start 2024-03-22 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Heavy drinking episodes | assessed at baseline and 3-month follow-up
  Number of past-month heavy drinking episodes (consuming 4+ drinks for females and 5+ drinks for males in one occasion)
Alcohol-related negative consequences | assessed at baseline and 3-month follow-up
  Number of alcohol-related negative consequences experienced in the past month

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Rowland, MA, Principal Investigator — Boston University Charles River Campus
Locations (1):
- Boston University Charles River Campus, Boston, Massachusetts, United States